CLINICAL TRIAL: NCT03781635
Title: Comparison of BIS Index Variations When i.v. Low-dose Ketamine is Administered Intraoperatively as Bolus Versus Continuous Infusion and Impact on the Anesthesia Gas Consumption.
Brief Title: Comparison of BIS Index Variations: Bolus Versus Infusion Ketamine, and Impact on the Anesthesia Gas Consumption
Acronym: KETABIS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Principal Investigator, Philippe Richebe, MD, PhD, Professor, Director of Research, Department of Anesthesiology and Pain Medicine of Maisonneuve-Rosemont Hospital, CIUSSS de l'Est de l'Ile de Montreal (CEMTL), Ciusss de L'Est de l'Île de Montréal
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018-1482
Record Dates: First submitted 2018-11-30; First posted 2018-12-20 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: Bolus Versus Infusion Ketamine, Anesthesia Gas Consumption
Keywords: Ketamine; anesthesia; BIS monitoring; epidural; intraoperative

STUDY DESIGN:
Intervention Model Description: Two groups of patients. Randomization into group infusion versus boluses of ketamine according to a randomization list for a total number of patients of 50.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization into group infusion versus boluses of ketamine will be done prior to the entrance in the OR, the day of the surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- bolus of intravenous ketamine (Active Comparator): A bolus of 0.25mg.kg-1 of ketamine will be first administered at the time of incision (T0) then every single hour for the rest of the surgery. Study starts at incision (T0) for ketamine administration and ends when the surgical team starts closing the deep layers of the abdominal incision.
  Interventions: Drug: bolus of intravenous ketamine
- continuous infusion of intravenous ketamine (Experimental): An infusion of 0.25 mg.kg-1.h-1 is started at T0 (incision) with an infusion pump and is kept at the same rate until the surgical team starts closing the deep layers of the abdominal incision. Consumption of the infusion pump is noted at T0 (incision) and at each hour during the surgery until the infusion is discontinued.
  Interventions: Drug: continuous infusion of intravenous ketamine

INTERVENTIONS:
Drug: bolus of intravenous ketamine — low-dose ketamine (0.25mg.kg-1) is administered intraoperatively as bolus at incision (T0) and for each hour of anesthesia untel the end of surgery.
  Arms: bolus of intravenous ketamine
Drug: continuous infusion of intravenous ketamine — An infusion of low-dose ketamine (0.25 mg.kg-1.h-1) is started at T0 (incision) with an infusion pump and is kept at the same rate until the end of surgery
  Arms: continuous infusion of intravenous ketamine

SUMMARY:
The aim of the present study is to show that i.v. ketamine boluses might lead to significant and clinically relevant BIS index increase that might lead to an increase in anesthesia dosing (halogenous gas) when compared to an i.v. continuous infusion of ketamine without any bolus.

DETAILED DESCRIPTION:
Hypothesis: The investigators hypothesize that BIS will not vary when ketamine is given as an i.v. infusion whereas BIS index will significantly vary when ketamine is given as intraoperative repeated bolus on an hourly basis. As a consequence, the bolus group might have a higher consumption of halogenous gases to keep BIS within normal values during anesthesia.

Background: ketamine is a pure NMDA-receptor antagonist widely used in anesthesia for its anesthetic and analgesic properties. However, boluses of intravenous ketamine have been reported to increase BIS values. The present study is the first to compare ketamine effect on BIS values when given as an infusion versus repeated boluses.

Objectives: primary objective: to measure the changes in BIS index values (delta BIS) after each bolus of i.v. ketamine 0.25mg.kg-1 given during anesthesia for surgeries lasting more than 3hs, and to demonstrate a significant increase of this BIS index whereas no significant increase is expected when i.v. ketamine is given as a continuous infusion intraoperatively. Secondary objectives: to measure the changes of BIS index values area under the curve when an infusion of i.v. ketamine 0.25mg.kg-1.h-1 is administered to the patient instead of boluses; to evaluate the time in minutes for the BIS index values to return within +/-10% of the pre-bolus values of this BIS index; to evaluate the time in seconds at which the peak of BIS will occur after ketamine bolus; to evaluate the consumption of halogenous gases during the entire surgery and for each hour of anesthesia (T0 = incision = time for first bolus of ketamine or start of ketamine infusion); to evaluate hemodynamic data (all the data from the ventilator and the monitor are recorded and exported per second) in both groups and see if the infusion group shows less hypotension events needing treatment with i.v. phenylephrine to stay within +/-20% of the mean blood pressure baseline; to evaluate the time for awakening, time for extubation, time spent in post-anesthesia care unit (PACU), delirium and cognitive functions in PACU (CAMshort assessment and MOCA).

Methods: REB from CR-HMR will be obtained. 50 patients undergoing elective general, urological, gynecological surgeries will be explained the study at the pre-anesthesia consultation and then fully consented the day of the surgery. Anesthesia protocol will be fully standardized in both the groups. BIS monitoring will be installed before induction of general anesthesia as well as the standard anesthesia monitoring. Randomization into group infusion versus boluses of ketamine will be done prior to the entrance in the OR, the day of the surgery. Ketamine will be given as follows: in the i.v. ketamine infusion group, an infusion of 0.25 mg.kg-1.h-1 is started with an infusion pump and is kept at the same rate until the surgical team starts closing the deep layers of the abdominal incision. Consumption of the infusion pump is noted at T0 (incision) and at each hour during the surgery and when the infusion is discontinued. In the i.v. ketamine bolus group, 0.25mg.kg-1 of ketamine will be first administered at the time of incision (T0) then every single hour for the rest of the surgery. Study starts at anesthesia induction and incision (T0) for ketamine administration and ends when the patient leaves the PACU. Objectives of the study are cited above.

Data analysis: statistical analyses will be done using SAS version 9.4 or higher and will be performed at a two-sided 0.05 significance level.

Significance/Importance: This is the first study that will compare the impact of the classical intraoperative ketamine administered as repeated i.v. boluses versus as a continuous i.v. infusion during major surgeries lasting more than 3 hours.

Study Design: open label study, with two controlled randomized parallel groups

Subject Population: ASA 1 to 3 adult patients scheduled to undergo elective general, urologic or gynecological surgeries.

Sample Size: 50 patients will be evaluated in this study.

Study Duration: 10 months.

Study Center: Maisonneuve-Rosemont Hospital, CIUSSS de l'Est de l'Ile de Montreal, Montreal, Quebec, Canada.

Adverse Events: None expected.

ELIGIBILITY:
Inclusion Criteria:

* ASA I to III
* Patients above 18yo
* Gender female or male
* Abdominal general, urological or gynecological surgery with epidural placement

Exclusion Criteria:

* BMI <18 or >35
* Chronic neurological or psychiatric disorder or history of stroke
* Use of psychotropic drugs within 2 weeks prior surgery
* Allergy to ketamine or its excipients or any drug of the anesthesia protocol of this study
* Any contra-indication or patient's refusal for epidural placement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of the increase of the BIS index (absolute value between 0 to 100) after each intravenous ketamine bolus | Intraoperative, during anesthesia
  To demonstrate and quantify à significant increase of the BIS index after each bolus of 0.25 mg.kg-1 ketamine given during surgeries lasting 3 hours and more, compared to an equivalent dose of ketamine given as a continuous infusion. Boluses of ketamine will start at T0 = incision and then will be repeated every hour for the duration of the surgery.

SECONDARY OUTCOMES:
Area under the curve of BIS values from T0=incision until end of the anesthesia, value without unit (area under curve) | Intraoperative, during anesthesia
  To compare the BIS index values area under the curve from T0=incision until end of anesthesia when i.v. ketamine 0.25mg.kg-1.h-1 is administered as an infusion or as hourly boluses.
Time for BIS to return within 10% of the baseline values (in minutes) | Intraoperative, during anesthesia
  To evaluate the time in minutes for the BIS index values to return within +/-10% of the values the BIS index had before the bolus of ketamine.
Time to reach the peak of BIS index after intravenous bolus of ketamine | Intraoperative, during anesthesia
  To evaluate the time in seconds at which the peak of BIS will occur after intravenous ketamine bolus 0.25mg/kg.
Evaluation of the consumption of halogenous gases (desflurane) during each hour of anesthesia in ml/kg/h of gas | Intraoperative, during anesthesia
  To evaluate the consumption of halogenous gases (desflurane) during each hour of anesthesia in ml/kg/h.
Evaluation of the consumption of phenylephrine in mcg/kg/h for each hour of anesthesia. | Intraoperative, during anesthesia
  To evaluate the need of intravenous phenylephrine given during each hour of anesthesia in both groups.
Evaluation of the blood pressure during each hour of anesthesia. | Intraoperative, during anesthesia
  To evaluate blood pressure recorded electronically during the whole anesthesia and to evaluate the impact of intravenous bolus of ketamine 0.25mg/kg on blood pressure during the whole hour following each bolus administration (given hourly).
Evaluation of the time in minutes necessary to extubatne the patient at the end of the surgery | End of surgery
  To evaluate the time for extubation in minutes at the end of surgery
Evaluation of the time in minutes to reach an Alerte score of >9 in post-anesthesia care unit | In post anesthesia care unit, 2 hours after surgery is done
  To evaluate the time in minutes to reach an alerte score (this score has no unit) of more than 9.
Evaluation of the MOCA score (score from 0 to 30) in PACU at 15 minutes after arrival in PACU (post-anesthesia care unit) | 15 minutes after arrival in PACU
  To evaluate the MOCA score (0 to 30) in PACU at 15minutes after arrival.
Evaluation of the MOCA score (score from 0 to 30) in PACU at 45 minutes after arrival in PACU (post-anesthesia care unit) | 45 minutes after arrival in PACU
  To evaluate the MOCA score (0 to 30) in PACU at 45minutes after arrival.
Evaluation of the delirium with CAM (Confusion Assessment Method that has NO unit) in PACU at 15 minutes after arrival in PACU (post-anesthesia care unit) | 15 minutes after arrival in PACU
  To evaluate the CAM (no unit) in PACU at 15minutes after arrival.
Evaluation of the delirium with CAM (Confusion Assessment Method that has NO unit) in PACU at 45 minutes after arrival in PACU (post-anesthesia care unit) | 45 minutes after arrival in PACU
  To evaluate the CAM (no unit) in PACU at 45minutes after arrival.
Evaluation of the total time spent in PACU in minutes | 3 hours after surgery
  Total time in PACU in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Philippe PR Richebé, MD PhD, Principal Investigator — CIUSSS Est de l'ile de Montreal
Locations (1):
- Hopital Maisonneuve Rosemont, CIUSSS de l'Est de l'Ile de Montreal, Montreal East, Quebec, Canada

REFERENCES:
- [Derived] Carrara L, Nault M, Morisson L, Godin N, Idrissi M, Fortier A, Guertin MC, Brulotte V, Fortier LP, Verdonck O, Richebe P. The impact of bolus versus continuous infusion of intravenous ketamine on bispectral index variations and desflurane administration during major surgery: The KETABIS study. Eur J Anaesthesiol. 2021 Nov 1;38(11):1168-1179. doi: 10.1097/EJA.0000000000001588. PMID 34474441